CLINICAL TRIAL: NCT06267885
Title: Fixation of Fracture Neck of Femur in Children by Cannulated Screws VS Wagner's Technique.
Brief Title: Fixation of Fracture Neck of Femur in Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mina Maged, Resident in assiut university hospital , orthopaedic department, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Children NOF fracture fixation
Record Dates: First submitted 2024-01-13; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Fracture Neck of Femur
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with fracture neck of femur fixed by cannulated screws (Active Comparator): Fix the fracture by two to three cannulatef screws
  Interventions: Procedure: Cannulated screws vs wagner's technique
- Patient with fracture neck of femur fixed by wagner's technique (Active Comparator): Fix the fracture by three to four k-wires
  Interventions: Procedure: Cannulated screws vs wagner's technique

INTERVENTIONS:
Procedure: Cannulated screws vs wagner's technique — Fixation of fracture neck of femur by cannulated screws or wagner's technique

SUMMARY:
Find the best way for fixation of fracture neck of femur in children either by cannulated screws or wagner's technique

DETAILED DESCRIPTION:
In the pediatric population, fracture of the neck of femur is relatively uncommon usually caused by high-energy trauma, but with high complication rates, despite appropriate diagnosis and management. The high rate of complication is due to the vascular anatomy of proximal femur.

Fracture neck of femur can be classified into transphyseal , transcervical (which is commonest), basal and pertrochanteric.

Complications include avascular necrosis, delayed union and non-union. Multiple fracture fixation methods have been used, with the overall goal being anatomic reduction with stable fixation.

Methods of fixation vary based on age, Delbet classification and dispalcement of the fracture.

Two types of fixation of pediatric fracture NOF of interest are cannulated screw (CS) and the Wagner technique.

Most studies agree that 3 screws are enough, and they should be inserted parallel in triangular arrangement with an inverted triangle. The CS should apply compression to the fracture (compression screws) to minimize the remaining fracture gap and accelerate the healing process. The use of washers allows for higher compression forces and thus increases the initial stabilization. CS shouldn't pass the physis in pediatrics to allow normal continuation of growth in children. The stability of fixation by CS has been shown to be affected by several factors: screw type, number, thickness, position and direction. Some of CS disadvantages are that they are mechanically unstable, failure of stabilization leads to varus malunion and it may lead to slipped capital femora epiphysis (SCFE) above the tips of the screws(especially short working distance in transcervical fractures).

The Wagner technique consists of the use of two or three k-wires bent as close as possible to the shaft and fixed to the shaft by two cerclage wires. Some advantages of this method are that k-wires can cross the physis and give good stability to the fracture with normal continuation of growth(especially in transphyseal & transcerviacal fractures). Hip spica is recommended to give more stabilization to the fixation and neutralize forces around the fixed fracture.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of fracture neck of femur
* children with age less than 14 years old

Exclusion Criteria:

* pathological fracture
* patients with cerebral palsy
* Associated ipsilateral femoral shaft fracture
* comminuted fractures
* old fracture ( > 2 weeks)

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
The better method for fixation of fracture neck of femur | Baseline, one year
  The rate of cases with complications with avascular necrosis in each method

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt